CLINICAL TRIAL: NCT07313358
Title: 10119473 -VIROMARKERS HDV Biomarkers Study
Status: Not yet recruiting | Type: Observational
Sponsor: University of Rome Tor Vergata (Other)
Collaborators: Euresist Network GEIE (Other); Informapro Srl (Other); Royal Free and University College Medical School (Other); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); EUROPEAN LIVER PATIENTS ASSOCIATION (Unknown)
Responsible Party: Principal Investigator, Valentina Svicher, Professor, University of Rome Tor Vergata
Other Study IDs: 101194735-HDV
Record Dates: First submitted 2025-11-25; First posted 2025-12-31 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: HDV Infection
Keywords: HDV infection; bulevirtide; biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — blood samples for testing of levels of HBsAg isoforms, HDV genotypes/subgenotypes and Altona/Qiagen HDV RNA quantification.
  The virological status of all participants enrolled will be assessed every 3 months, according to the guidelines promoted by European Association for the Study of the Liver in 2023, at week 48, 96 and 144 after enrollment. The 48-, 96- and 144-week follow-up status assessment will include:
  HDV RNA levels ALT levels Adverse events Liver-related events Hospitalization, including length of stay The use of stored specimens will be reviewed and approved by the Protocol Team, the VIROMARKERS Scientific Steering Committee, and EC Horizon Europe.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- HDV-BLV: patients with HDV infection who initiated BLV from January 2023 to February 2025 for whom retrospective data and samples are available. Follow-up and sample collection will be extended for this population over the period of the study grant.
  To be eligible for inclusion in both the retrospective and prospective part of the study, participants have to be ≥18 years of age, have signed an informed consent and satisfy the following additional criteria:
  A diagnosis of chronic HDV infection with or without compensated cirrhosis Having started BLV monotherapy 2mg/day according to the criteria reported in the recent clinical practice guidelines on HDV infection promoted by EASL [EASL CPG 2024] Be under effective treatment with nucleoside analogues with HBV-DNA <20 IU/ml at the time of starting BLV

SUMMARY:
This is an observational study, in which clinical data, samples, and any other procedures possibly already performed on participants, were performed within the scope of clinical practice or within the scope of otherwise authorized projects, and that therefore there are no procedures performed specifically for this study, which instead uses data collected previously or prospectively during an extended follow-up, but in any case within the scope of current clinical practice. Most participants have been enrolled and followed up at the project partners' clinical sites over 2023-2025. Their follow-up and sample collection will continue over the duration of the project. At the time of enrollment, demographics, medical history, medications and treatments prescribed were recorded and will be used in this study if the participant consent to be included also in VIROMARKERS. HDV genotypes/subgenotypes will be determined ex-novo on existing baseline stored samples.

The harmonization of HDV-RNA assays by utilizing standardized and validated flowcharts still represents a relevant diagnostic unmet clinical need for the appropriate monitoring of patients with CHD receiving BLV treatment. Furthermore, information on long-term virological response and factors predictive of virological outcome is scarce.

Specific primary objectives to characterise the response to bulevirtide in CHD include:

* To estimate the percentage of participants who will achieve virological response (defined as a decline in serum HDV RNA of >2 log or to undetectable HDV-RNA) and the proportion achieving undetectable HDV-RNA at week 48, 96 and 144 weeks of BLV treatment.
* To estimate the percentage of participants who will achieve biochemical response and combined response (defined as achievement of virological response and ALT normalization) at week 48, 96 and 144 weeks of BLV treatment.
* To evaluate whether HDV-RNA levels at baseline or their kinetics during the first 12 weeks of BLV treatment can predict the achievement of undetectable serum HDV-RNA during BLV treatment.

DETAILED DESCRIPTION:
For each participant, a blood sample was obtained at baseline and every 3 months during BLV treatment up to week 96. For a subset of participants, blood samples collected up to 144 weeks of treatment will be also available for analysis. At each time point, serum HDV-RNA was quantified with the reference RoboGene 2.0 assay used in clinical studies aimed at evaluating the efficacy of BLV.

For a subset of 80 participants followed-up at the Infectious Disease and Hepatology Unit of the University of Rome Tor Vergata and at the Policlinico of Milano, HDV RNA quantification using Altona (AltoStar assays), Qiagen and RoboGene 2.0 will be performed retrospectively in samples stored in 2023-2025 as well as in newly collected samples in 2025-2028. This will allow a comparison of the diagnostic performances of these assays and their capability to predict the achievement of virological response or undetectable HDV-RNA at week 48 and 96 and at week 144 in a subset. As such for the association analysis it will be conducted separate analyses according to the method of quantification used. Particular attention will be dedicated at comparing the sensitivity of the above-mentioned assays by evaluating their ability to detect residual HDV viremia during treatment.

Also, on this subset of approximately 80 individuals, the levels of the three different isoforms of HBsAg (L-, M- and S-HBs) will be quantified by using three different ad-hoc designed ELISA assays at the following time points: baseline, 48, and 96 weeks and 144 weeks for selected patients. These assays have been demonstrated to have high sensitivity (detection limit for each protein is 0.1 ng/ml) and a high specificity, taking advantage of a sandwich system based on anti-PreS1, anti-PreS2 and anti-S antibodies, respectively. For each patient and for each time point, total HBsAg, L-HBs, M-HBs and S-HBs levels will be quantified in duplicate.

In the analysis, the virological status of each participant enrolled will be assessed every 3 months according to the guidelines promoted by European Association for the Study of the Liver and up to 144 weeks.

The use of stored clinical specimens within this protocol will be reviewed by the Protocol Team, the VIROMARKERS Scientific Steering Committee, and EC Horizon Europe.

Specific secondary objectives include comparing the diagnostic performances of available assays for HDV-RNA quantification; comparing the rates of undetectable serum HDV-RNA at week 48, 96 and 144 by different HDV-RNA assays; comparing the kinetics of HDV-RNA during BLV treatment by different assays for HDV-RNA quantification; evaluating if the levels of HBsAg isoforms, alone or in combination with serum HDV-RNA at baseline, can predict the achievement of virological response to BLV at at week 48, 96 and 144 and comparing the rate of virological response to BLV according to HDV genotypes/subgenotypes.

The information used from this study on participants with CHD will be rapidly analyzed and shared broadly to guide policymakers for the use and monitoring of response to BLV and to design future studies.

Participant Selection The study will include 220 patients who initiated BLV from January 2023 to February 2025 for whom retrospective data and samples are available. Follow-up and sample collection will be extended for this population over the period of the study grant.

To be eligible for inclusion in both the retrospective and prospective part of the study, participants have to be ≥18 years of age, have signed an informed consent and satisfy the following additional criteria:

A diagnosis of chronic HDV infection with or without compensated cirrhosis Having started BLV monotherapy 2mg/day according to the criteria reported in the recent clinical practice guidelines on HDV infection promoted by EASL Be under effective treatment with nucleoside analogues with HBV-DNA <20 IU/ml at the time of starting BLV

Study Design This is a mainly retrospective and partly prospective observational study which will enrol patients with CHD who started BLV over 2023- March 2025. Participants were enrolled in other projects and most have already been followed for some time as part of these studies and will be enrolled in this new study at the time of signing the consent to participate in VIROMARKERS.

Participants have been followed for a minimum of 96 weeks for achievement of virological response. Similar inclusion criteria and follow-up with additional sample collection and testing (levels of HBsAg isoforms, HDV genotypes/sub genotypes) are planned for the prospective part which encompasses an extension of follow-up for those already recruited in the retrospective phase. No new enrolments are planned for this protocol.

Study Objectives Primary and secondary objectives are listed below.

Primary Characterize individuals with CHD in terms of demographics, co-morbidities and HDV disease status Describe the virological and clinical course under treatment with BLV for all participants Estimate the proportion of participants achieving a virological response (defined as a decline in serum HDV RNA of >2 log or undetectable HDV-RNA) and undetectable HDV-RNA by 48, 96, 144 weeks from starting BLV Estimate the percentage of patients who achieve biochemical response and combined response (defined as achievement of virological response and ALT normalization) at 48, 96, 144 weeks from starting BLV Identify potential predictors of response: HDV-RNA levels at baseline, HDV-RNA kinetics during the first 12 weeks In a subset of the study population, to measure levels of HBsAg isoforms, along or in combination with serum HDV-RNA at baseline and over follow-up and HDV genotypes/subgenotypes at baseline.

Secondary In a subset of the study population with multiple measures, to compare the diagnostic performances of the assays for HDV-RNA quantification by Robogene, Altona (AltoStar assays) and Qiagen, against the WHO reference standard and clinical samples with known serum HDV RNA.

To trace and compare the kinetics of HDV-RNA during BLV treatment by using different assays for HDV-RNA quantification.

To compare the rate of undetectable serum HDV-RNA up to 144 weeks by different assays for HDV-RNA quantification.

Sample Size Sample size for the retrospective part was closed at 220 individuals. Are expected further recruitments over the 3 years of the grant. It is uncertain how many participants will start treatment each year. With the infrastructure that is in place, recruitment of patents in need for treatment will be rapid although it is a rare disease, so the forecast is to further enroll a maximum of 30 additional individuals.

Based on the population of individuals previously studied and who can be potentially enrolled and follow-ed up in VIROMARKERS, the expectation is to have a study population with a median age of 50 years (range 30-70) with a comparable gender distribution, 95% of European origin. Sites in diverse geographic locations in several countries have participated. By contrast, the prospective samples will be collected only in Italy at the project sites in Policlinico University of Milan and Rome (University of Tor Vergata).

For CHD participants on BLV, data from a single trial exist to estimate the percentage of participants who will achieve virological response by week 48 and to determine power for studying risk factors related to response.

Statistical considerations are summarized below. In the study are considered binary as well continuous predictors, e.g., HDV RNA, HDV RNA slope, etc.). For the latter, power was estimated from comparing the upper versus lowest quartile of the factor.

In a recent analysis of 244 persons with CHD in the SAVE-D study, 48% achieved undetectable HDV-RNA and 79% virological response. Using these data, relative risks of 2.21 and 2.50 can be detected with 80% and 90% power, respectively, assuming 100 participants will achieve undetectable serum HDV-RNA). For virological response and ALT normalization which have higher response rates, the power will be greater. We expect to have HBsAg isoforms measured in a subset of 80 individuals, so the power will be limited for this analysis for ORs in the range of 1.8-2.8, depending on the rate of enrolment of new initiators.

Participant Selection Inclusion Criteria

To be eligible for enrollment participants must:

Be > 18 years of age Sign an informed consent Have a diagnosis of HDV infection with or without compensated cirrhosis Having started BLV monotherapy 2mg/day according to the criteria reported in the recent clinical practice guidelines on HDV infection promoted by EASL in 2023.

Be under effective treatment with nucleoside analogues with HBV-DNA <20 IU/ml at the time of starting BLV Exclusion Criteria Decompensated liver disease BLV combined with pegIFN Past treatment with BLV

ELIGIBILITY:
Inclusion Criteria:

* Be > 18 years of age
* Sign an informed consent
* Have a diagnosis of HDV infection with or without compensated cirrhosis
* Having started BLV monotherapy 2mg/day according to the criteria reported in the recent clinical practice guidelines on HDV infection promoted by EASL (EASL CPG 2023)
* Be under effective treatment with nucleoside analogues with HBV-DNA <20 IU/ml at the time of starting BLV

Exclusion Criteria:

* Decompensated liver disease
* BLV combined with pegIFN
* Past treatment with BLV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: participants have to be ≥18 years of age, have signed an informed consent and satisfy the following additional criteria: A diagnosis of chronic HDV infection with or without compensated cirrhosis Having started BLV monotherapy 2mg/day according to the criteria reported in the recent clinical practice guidelines on HDV infection promoted by EASL [EASL CPG 2024] Be under effective treatment with nucleoside analogues with HBV-DNA <20 IU/ml at the time of starting BLV
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
HDV Viral Load | 48, 96, 144 weeks after starting Bulevirtide
  HDV-RNA decline > 2 log OR reaching undetectable HDV-RNA

CONTACTS AND LOCATIONS:
Overall Officials: PIETRO LAMPERTICO, PROFESSOR, Principal Investigator — UNIVERSITA' DI MILANO
Locations (2):
- Heinrich Heine University, Düsseldorf, Germany, Germany
- Università di Milano, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: Yes
The access to the data, both for view, upload and download will be monitored with "Access control logging", based on a user authentication control with geolocalization of the access, based, for example, on Google authenticated accounts - Google Workspace or similar.
  The repository of the database will be located on the INFORMAPRO/EURESIST organization Google WorkSpace Shared Drive infrastructure, located in the EU space, as the organizations are Italian and by contract, the hosted workspace is inside the EU space.
  In order to make the data interoperable, it is important to have 3 basic features:
  A STANDARDIZED Metadata. This standardization has to be developed with the common efforts of all WP participated partners
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Start date: july 31 2025 end dat: not defined
Access Criteria: Any researcher can apply for the access to the Project Coordinator
URL: https://www.viromarkers.eu/

REFERENCES:
- [Background] Rodgers MA, Shah PA, Anderson M, Vallari AS, Gersch J, Mbanya D, Sauleda Oliveras S, Choudhry S, Leary TP, Kuhns MC, Dawson GJ, Cloherty GA, Lau DTY. Characterization of HBV surface antigen isoforms in the natural history and treatment of HBV infection. Hepatol Commun. 2023 Apr 4;7(4):e0027. doi: 10.1097/HC9.0000000000000027. eCollection 2023 Apr 1. PMID 37026760
- [Background] Charre C, Regue H, Deny P, Josset L, Chemin I, Zoulim F, Scholtes C. Improved hepatitis delta virus genome characterization by single molecule full-length genome sequencing combined with VIRiONT pipeline. J Med Virol. 2023 Mar;95(3):e28634. doi: 10.1002/jmv.28634. PMID 36879535
- [Background] Pfefferkorn M, Bohm S, Schott T, Deichsel D, Bremer CM, Schroder K, Gerlich WH, Glebe D, Berg T, van Bommel F. Quantification of large and middle proteins of hepatitis B virus surface antigen (HBsAg) as a novel tool for the identification of inactive HBV carriers. Gut. 2018 Nov;67(11):2045-2053. doi: 10.1136/gutjnl-2017-313811. Epub 2017 Sep 26. PMID 28951526
- [Background] Wedemeyer H, Aleman S, Brunetto MR, Blank A, Andreone P, Bogomolov P, Chulanov V, Mamonova N, Geyvandova N, Morozov V, Sagalova O, Stepanova T, Berger A, Manuilov D, Suri V, An Q, Da B, Flaherty J, Osinusi A, Liu Y, Merle U, Schulze Zur Wiesch J, Zeuzem S, Ciesek S, Cornberg M, Lampertico P; MYR 301 Study Group. A Phase 3, Randomized Trial of Bulevirtide in Chronic Hepatitis D. N Engl J Med. 2023 Jul 6;389(1):22-32. doi: 10.1056/NEJMoa2213429. Epub 2023 Jun 22. PMID 37345876
- [Background] Brancaccio G, Salpini R, Piermatteo L, Surdo M, Fini V, Colagrossi L, Cantone M, Battisti A, Oda Y, Di Carlo D, Ceccherini-Silberstein F, Perno CF, Gaeta GB, Svicher V. An Increase in the Levels of Middle Surface Antigen Characterizes Patients Developing HBV-Driven Liver Cancer Despite Prolonged Virological Suppression. Microorganisms. 2021 Apr 2;9(4):752. doi: 10.3390/microorganisms9040752. PMID 33918474
- [Background] Stelzl E, Ciesek S, Cornberg M, Maasoumy B, Heim A, Chudy M, Olivero A, Miklau FN, Nickel A, Reinhardt A, Dietzsch M, Kessler HH. Reliable quantification of plasma HDV RNA is of paramount importance for treatment monitoring: A European multicenter study. J Clin Virol. 2021 Sep;142:104932. doi: 10.1016/j.jcv.2021.104932. Epub 2021 Jul 24. PMID 34333392
- [Background] Degasperi E, Anolli MP, Jachs M, Reiberger T, De Ledinghen V, Metivier S, D'Offizi G, di Maria F, Schramm C, Schmidt H, Zollner C, Tacke F, Dietz-Fricke C, Wedemeyer H, Papatheodoridi M, Papatheodoridis G, Carey I, Agarwal K, Van Bommel F, Brunetto MR, Cardoso M, Verucchi G, Ciancio A, Zoulim F, Aleman S, Semmo N, Mangia A, Hilleret MN, Merle U, Santantonio TA, Coppola N, Pellicelli A, Roche B, Causse X, D'Alteroche L, Dumortier J, Ganne N, Heluwaert F, Ollivier I, Roulot D, Vigano M, Loglio A, Federico A, Pileri F, Maracci M, Tonnini M, Arpurt JP, Barange K, Billaud E, Pol S, Gervais A, Minello A, Rosa I, Puoti M, Lampertico P. Real-world effectiveness and safety of bulevirtide monotherapy for up to 96 weeks in patients with HDV-related cirrhosis. J Hepatol. 2025 Jun;82(6):1012-1022. doi: 10.1016/j.jhep.2024.12.044. Epub 2025 Jan 8. PMID 39793613
- See also: Related Info — https://www.viromarkers.eu/

DOCUMENTS (1):
  • Study Protocol (2025-04-30): https://cdn.clinicaltrials.gov/large-docs/58/NCT07313358/Prot_000.pdf